CLINICAL TRIAL: NCT03583645
Title: Prevention of Aggressive Behavior in Adolescents by Means of an Intervention Based on Implicit Theories of Personality
Brief Title: The Effect of an Intervention Based on Implicit Theories of Personality on the Prevention of Adolescent Dating Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Medikosta IMQ Análisis Clínicos (Unknown)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI_2016_1_0023
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Dating Violence
Keywords: Adolescence; Prevention; Aggressive behavior; Dating Violence
MeSH Terms: conditions — Aggression | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio blocked by gender to one of two groups: experimental condition (ITP intervention) versus control condition (educational intervention) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation was concealed to the participants, researchers -who were in class the assessment days- and teachers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental theory of personality (Experimental): 1 hour behavioral intervention (based on ITP) consisting on several tasks to be completed on paper individually.
  Interventions: Behavioral: Incremental theory of personality
- Educational intervention (Other): 1 hour educational intervention (about the human brain) consisting on several tasks to be completed on paper individually.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Behavioral: Incremental theory of personality — The experimental intervention (originally developed by David S. Yeager and colleagues) teaches that individuals have the potential to change. It has three main parts. First, participants are asked to read scientific studies that provide evidence that behaviors are controlled by "thoughts and feelings in brains," and that pathways in the brain have the potential to be changed under the right circumstances. Second, participants read several testimonials purportedly written by upperclassmen to bring credibility to the ITP. Finally, participants are asked to write their own version of such a narrative. This self-persuasive writing exercise has been shown to facilitate the internalization of the intervention message, building on a long line of research on cognitive dissonance.
  Arms: Incremental theory of personality
Other: Educational Intervention — The educational intervention involved scientific information about the human brain. It was designed to be parallel to the experimental intervention and, hence, it has also three main parts. First, participants are asked to read scientific information about the different areas of the brain and their specialties. Second, participants read several testimonials written by upperclassmen about their transition to high school and how their brains help them to adapt to the new space and all the physical differences of the building and the classes. Finally, participants are asked to write a letter to another student explaining the main things he or she has learned about the brain and thinks are important for adapting to the new physical environment in high school.
  Arms: Educational intervention

SUMMARY:
This study evaluates the efficacy of an intervention based on the Implicit Theories of Personality (ITP) to prevent dating violence in Spanish adolescents. Half of participants received the ITP intervention, while the other half received an educational intervention.

DETAILED DESCRIPTION:
Intimate partner violence is a problem arising in adolescence, which causes severe suffering. Since the first romantic relationships are established during adolescence, implementation of preventive interventions during this developmental stage opens a window of opportunity for the prevention of partner aggression. Previous prevention programs have shown efficacy in modifying cognitions and attitudes related to dating violence, although behavioral changes have been reported in very few cases. Recent innovative brief interventions based on changing entity theories of personality (i.e., the belief that people cannot change and personal characteristics are fixed; Miu & Yeager, 2015) have provided good results for preventing depression and other behavioral problems in adolescents. Therefore, the principal aim of this study is to examine whether a brief one-hour intervention based on promoting the idea that people can change shows efficacy in the prevention of perpetration and victimization of dating aggressive behaviors (both online -cyber dating abuse- and traditional -face-to-face dating aggression-) in adolescents. Additionally, other objective of the project is to examine whether gender moderates the effects of the intervention in changes in dating violence. The study involves the evaluation of the intervention in a sample of around 400 adolescents (13-18 years), randomly allocated to experimental and control conditions. It is a field experiment conducted in high schools and involves multiple measures over time (self-reports and parent reports). In summary, the project aims to respond to the challenge of health and wellness in the population through a randomized controlled trial with multiple sources of measure and from a biopsychosocial perspective. The ITP intervention has the potential to become a universal intervention to help reduce the rates of adolescent dating violence.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the adolescents and their parents.
* To be fluent in Spanish.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 402 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores of the Dating Violence Questionaire (developed by the research team) at 2 weeks, 6 months, and 12 months. | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported dating aggressive behaviors during the last 6 months (last week in the 1 week follow-up) measured by 25 items scored 0-3 (0 = never; 3 = often), yielding a total between 0 and 75.

OTHER OUTCOMES:
Affection and Communication subscale of the Parenting Style Scale (Oliva, Parra, Sanchez-Queija, & López, 2007) for parents. | Baseline and 6 months.
  8 items reported by the adolescents' parents from the affection and communication subscale, which assesses support and care delivered by the parents, their ability to be there, and the communication between them. Each item is scored 1-6 (1= not at all true to 6=completely true), yielding a total between 8 and 48.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be provided to the journals in which it is planned to publish the results of the study. In addition, the PI and research team will consider to make IPD available to other researchers after publishing the results of the study.

DOCUMENTS (2):
  • Informed Consent Form (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03583645/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03583645/Prot_SAP_003.pdf